CLINICAL TRIAL: NCT01707056
Title: The Effect of Coffee Consumption on the Intestinal Absorption of Levothyroxine Thyroid Hormone Replacement in Patients With Thyroid Carcinoma
Brief Title: The Effect of Coffee on the Absorption of Thyroid Hormone in Patients With Thyroid Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011-338
Record Dates: First submitted 2012-10-05; First posted 2012-10-15 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Carcinoma; Hypothyroidism
Keywords: levothyroxine; synthroid; coffee; absorption; tea; thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Hypothyroidism | interventions — Coffee; Milk; Tea; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Black coffee (Active Comparator): Synthroid will be administered with 12 ounces of black coffee for a period of 6 weeks.
  Interventions: Other: Black Coffee
- Coffee with Milk (Active Comparator): Synthroid will be administered with 12 ounces of coffee and 2 ounces of 2% milk for a period of 6 weeks.
  Interventions: Other: Coffee with Milk
- Black Tea (Active Comparator): Synthroid will be administered with 12 ounces of black Lipton tea for a period of 6 weeks.
  Interventions: Other: Black Tea
- Water (Placebo Comparator): Synthroid will be administered with 12 ounces of water for a period of 6 weeks.
  Interventions: Other: Water

INTERVENTIONS:
Other: Black Coffee — Taking Synthroid with 12 ounces of black coffee for 6 weeks.
  Arms: Black coffee
Other: Coffee with Milk — Taking Synthroid with 12 ounces of black coffee and 2 ounces of 2% milk for a period of 6 weeks.
  Arms: Coffee with Milk
Other: Black Tea — Taking Synthroid with 12 ounces of black tea for a period of 6 weeks.
  Arms: Black Tea
Other: Water — Taking Synthroid with water for a period of 6 weeks.
  Arms: Water

SUMMARY:
The purpose of this study is to evaluate whether taking thyroid hormone medication with beverages other than water, decreases absorption of the medication by the intestine. Specifically we are interested in whether coffee, coffee with milk, or black tea affects how thyroid medication is absorbed by the body. Previous studies have suggested that taking thyroid hormone with coffee may interfere with the ability to absorb thyroid medicine. Given that many patients take their thyroid medicine with beverages other than water, and specifically with coffee or tea, understanding whether and how much coffee or tea may decrease thyroid hormone absorption is important for clinical practice.

This study will help determine the safest and most effective way for adults to take their thyroid medication and will guide medical practitioners in how to counsel their patients when they prescribe thyroid hormone.

DETAILED DESCRIPTION:
Previous studies have suggested that taking thyroid replacement therapy with coffee potentially hinders its absorption. We already know that food especially a fiber-rich diet, cholestyramine resin, aluminum containing antacids, activated charcoal, and certain herbal remedies among others interfere with the ability to absorb thyroid medicine. These findings have prompted providers to advise patients to take their levothyroxine on an empty stomach in the morning. However, many patients take their thyroid medicine with their morning cup of coffee prior to eating breakfast. A small study has shown that Italian espresso coffee can decrease the absorption of levothyroxine, but the effect of American style coffee is not known. Given that the intestinal absorption of levothyroxine can be hindered by multiple substances and coffee is the most commonly consumed beverage worldwide, it is important to investigate what effect coffee may have on thyroid hormone absorption and thyroid function tests.

Using methods similar to those used in previous studies, this study will measure thyroid function tests in approximately 10-20 subjects (18-60 years of age) over a 6 hour period of time after taking their thyroid medication with the specified study beverage for a 6 week period. Subjects will be randomized to water, black coffee, coffee with milk, and black tea as four specified study beverages, with water serving as the control beverage. Each subject will be recruited to participate with each study beverage for a 6 week period of time in a total of four consecutive 6 week periods. Blood draws will occur at the end of each 6 week period on test days 1, 2, 3, and 4. The coffee will represent the most common household coffee brand, Folgers. Thyroid function tests with each beverage will be compared to thyroid function tests with water to determine if thyroid medication absorption is impaired by coffee, coffee with milk, or tea.

This study will help determine the safest and most efficacious way for adults to take their thyroid medication and will guide medical practitioners in how to counsel their patients when they prescribe thyroid replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

- patients with thyroid carcinoma after standard care of treatment on stable dose of Synthroid with a detectable baseline TSH

Exclusion Criteria:

* Pregnancy
* Undetectable baseline TSH
* Not willing to drink coffee, coffee with milk, or black tea
* Age less than 18 or greater than 60 years old
* Taking generic thyroid hormone (levothyroxine) and not brand-name Synthroid
* Dose of thyroid medication has been recently changed (less than 3 months ago)
* Currently receiving treatment for gastroesophageal reflux disease, gastritis, stomach or intestinal cancer, inflammatory bowel disease, or H. pylori
* Taking cholestyramine resin, colestipol hydrochloride, sucralfate, iron sulphate, aluminum containing antacids, activated charcoal, raloxifene, and herbal remedies
* History of previous gastric or small intestine surgery
* Diagnosis of kidney or liver disease, congestive heart failure, anemia, biliary disease, pancreatitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in TSH (thyrotropin-stimulating-hormone) with each beverage type | 6 hours
  1. change in TSH over 6 hours
  2. peak change in TSH over 6 hours

SECONDARY OUTCOMES:
Change in TSH with various beverages | 6 weeks
  To determine if taking Synthroid for 6 weeks with each of the prescribed study beverages results in a different baseline TSH, reflecting altered absorption of levothyroxine with each particular beverage.
Change in total T4 with each beverage type | 6 hours
  1. Change in total T4 over 6 hours
  2. Peak change in total T4 over 6 hours
  3. area under the curve (AUC) for total T4
Change in free T4 with each beverage type | 6 hours
  1. Change in free T4 over 6 hours
  2. Peak change in free T4 over 6 hours
  3. area under the curve (AUC) for free T4
Change in total T3 with each beverage type | 6 hours
  1. Change in total T3 over 6 hours
  2. Peak change in total T3 over 6 hours
  3. area under the curve (AUC) for total T3

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Krajewski, MD, Principal Investigator — MedStar Health
Locations (3):
- United States (3):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar St. Mary's Hospital, Leonardtown, Maryland

REFERENCES:
- [Background] Benvenga S, Bartolone L, Pappalardo MA, Russo A, Lapa D, Giorgianni G, Saraceno G, Trimarchi F. Altered intestinal absorption of L-thyroxine caused by coffee. Thyroid. 2008 Mar;18(3):293-301. doi: 10.1089/thy.2007.0222. PMID 18341376